CLINICAL TRIAL: NCT02759887
Title: Longitudinal Assessment of Amyloid Positron Emission Tomography (PET), Fludeoxyglucose F18 (FDG) PET, Tau PET, Magnetic Resonance Imaging (MRI), and Blood Spot Ribonucleic Acid (RNA) in Down Syndrome Individuals With and Without Alzheimer's Dementia and Normal Controls
Brief Title: Relationship Between Down Syndrome (DS) and Alzheimer's Disease (AD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Banner Alzheimer's Institute, Phoenix (Unknown); Translational Genomics Research Institute (TGEN), Phoenix (Unknown)
Responsible Party: Principal Investigator, Pam Dewey, Research Clinician, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PHX-16-0028-70-03
Record Dates: First submitted 2016-04-15; First posted 2016-05-03 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Down Syndrome; Alzheimer's Dementia
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease | interventions — Fluorodeoxyglucose F18; Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DS adult group (Other): Consists of 15 DS subjects aged 21 and older who do not qualify for the diagnosis of dementia at the beginning of the study. Interventions include biospecimen collection, cognitive assessments, caregiver questionnaire, Florbetapir F18 imaging, MRI, Fludeoxyglucose F18 (FDG), Tau Pet, Actigraphy.
  Interventions: Procedure: biospecimen collection; Other: cognitive assessments; Other: caregiver questionnaire; Procedure: Florbetapir F18 imaging; Procedure: MRI; Procedure: Fludeoxyglucose F18 (FDG); Procedure: Tau Pet; Procedure: Actigraphy
- DS/AD group (Other): Consists of 15 DS subjects aged 40 and older who do qualify for the diagnosis of dementia by DSM-IV criteria. Diagnoses will be by standard consensus review of all cases. Interventions include biospecimen collection, cognitive assessments, caregiver questionnaire, Florbetapir F18 imaging, MRI, Fludeoxyglucose F18 (FDG), Tau Pet, Actigraphy.
  Interventions: Procedure: biospecimen collection; Other: cognitive assessments; Other: caregiver questionnaire; Procedure: Florbetapir F18 imaging; Procedure: MRI; Procedure: Fludeoxyglucose F18 (FDG); Procedure: Tau Pet; Procedure: Actigraphy
- NC adult (Other): Consists of 10 cognitively normal, non-DS individuals, age-matched to the DS adult group. Interventions include biospecimen collection, cognitive assessments, Florbetapir F18 imaging, MRI, Fludeoxyglucose F18 (FDG), Tau Pet, Actigraphy.
  Interventions: Procedure: biospecimen collection; Other: cognitive assessments; Procedure: Florbetapir F18 imaging; Procedure: MRI; Procedure: Fludeoxyglucose F18 (FDG); Procedure: Tau Pet; Procedure: Actigraphy

INTERVENTIONS:
Procedure: biospecimen collection — Blood: ApoE genotyping, comprehensive metabolic panel, RNA sequencing. Urine: beta-hCG (human corionic gonadotropin) testing.
Other: cognitive assessments — Dementia Questionnaire for People with Learning Disabilities; Mini-Mental State Examination; Severe Impairment Battery; Vineland Adaptive Behavior Scale; Arizona Memory Assessment for Intellectual Disability; Kaufman Brief Intelligence Test; Nepsy Mazes; and, Timed Up and Go.
Other: caregiver questionnaire
  Arms: DS adult group; DS/AD group
Procedure: Florbetapir F18 imaging — Used in small doses to image brain amyloid-beta deposits in human beings. Radioactivity necessary to create the positron emission tomography (PET) images. Radiation exposure is slightly more than a person would receive from a routine clinical head computed tomography scan.
Procedure: MRI — Magnetic resonance imaging of the head and brain.
Procedure: Fludeoxyglucose F18 (FDG) — Injected intravenously during a PET scan and is a marker for the tissue uptake of glucose; a radiopharmaceutical compound.
Procedure: Tau Pet — Administered during a PET, in small amounts, necessary to create the scan images. Radioactive. The total amount of radiation is about the same that a patient receives from a routine abdominal/pelvis computerized tomography.
  Other Names: F-AV-1451
Procedure: Actigraphy — A non-invasive method of monitoring human rest and activity cycles. A small actigraph unit is worn to measure gross motor activity. The unit is usually worn on the wrist.
  Other Names: actimetry

SUMMARY:
In order to treat individuals with Down syndrome (DS) better and more efficiently and to gain more insights on its relation to Alzheimer's disease (AD), a comprehensive understanding is needed for its progression in the early or preclinical phase using various biomarkers. DS is a significant risk factor for the early development of AD, with plaques and tangles typically developing by age 35. A better understanding is needed of early markers of the disease in DS patients. Additionally the DS population represents a unique group - due to this elevated risk for AD - to examine biomarkers that may translate in general outside of the DS population to individuals at risk for developing late onset AD. In this proposal, the researchers will assess the longitudinal changes of various biomarkers in a cohort of individuals similar in design to the cross-sectional sectional study in the preliminary data.

DETAILED DESCRIPTION:
This study will recruit from three experimental groups: (1)The DS (adult) group will consist of 15 DS subjects aged 21 and older who do not qualify for the diagnosis of dementia at the beginning of the study. (2)The DS/AD group will consist of 15 DS subjects aged 40 and older who do qualify for the diagnosis of dementia by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria. Diagnoses will be by standard consensus review of all cases. (3)Normal control (NC) adult will consist of 10 cognitively normal, non-DS individuals, age-matched to the DS group. Blood will be collected to assess apolipoprotein E (ApoE) genotype. Participation in the dried blood spot collection (DBSC) will be an optional sub-study. Only participants and/or their caregivers/legally authorized representatives indicating they wish to have DBSC performed on the consent will provide specimens.

ELIGIBILITY:
Inclusion criteria for Non-AD/DS subjects:

* Subjects with free Trisomy 21.
* Male or female subjects who are 21 years of age or older.
* Subjects who are not diagnosed with possible or probable AD or dementia after evaluation NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke- Alzheimer's Disease and Related Disorders Association) criteria.
* Subjects who live with or have regular visits from a responsible caregiver willing to provide information about the subject's cognitive status.
* If the subject is incapable of giving informed consent, the caregiver may consent on behalf of the subject (subject must still confirm assent).

Inclusion criteria for AD/DS subjects:

* Subjects with free Trisomy 21.
* Male or female subjects who are 40 and older years of age.
* Subjects who are diagnosed with possible or probable using NINCDS-ADRDA criteria.
* Subjects who live with or have regular visits from a responsible caregiver willing to provide information about the subject's cognitive status.
* If the subject is incapable of giving informed consent, the caregiver may consent on behalf of the subject (subject must still confirm assent).

Inclusion criteria for Normal Controls

* Cognitively normal, non-DS individuals.
* Age-matched to the DS group.
* Subjects who signed an Institutional Review Board-approved informed consent.

Exclusion Criteria: (for all groups)

* Previous or current diagnosis of a neurodegenerative disorders other than AD or DS, including, but not limited to Parkinson's disease, Pick's disease, fronto-temporal dementia, Huntington's chorea, Creutzfeldt-Jacob disease, normal pressure hydrocephalus, and progressive supranuclear palsy.
* Previous or current diagnosis of other dementing/neurodegenerative disease (e.g. Parkinson's disease dementia, dementia with Lewy bodies, Lewy body variant AD).
* Previous or current diagnosis of mixed dementia.
* Previous or current diagnosis of cognitive impairment resulting from other known etiology.
* Previous or current diagnosis of clinically significant infarct or possible multi-infarct dementia as defined by the National Institute of Neurological Disorders and Stroke/Association Internationale pour la Recherche et l'Enseignement en Neuroscience (NINDS-AIREN) criteria.
* Previous or current evidence on screening MRI, computed tomography (CT), or other biomarker studies that suggests an alternate etiology (other than probable AD in patients with AD) for cognitive deficit; or in the case of non-AD controls any evidence on screening MRI, CT, or other biomarker studies that suggests the presence of AD pathology. Brain amyloid-β peptides (Aβ) on Amyloid imaging/PET imaging, however, is expected in many non-AD/DS and all AD/DS subjects, and will not be grounds for exclusion.
* Previous or current clinically significant psychiatric disease, as judged by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria, particularly current major depression or schizophrenia. Patients with dementia who are experiencing behavioral disturbances that may require treatment with psychotropic medications may be entered only after discussion and with the approval of the principal investigator. The investigators should carefully consider whether subjects with behavioral dysfunction will be able to complete the imaging session.
* Previous or current history of epilepsy or convulsions, except for febrile convulsions during childhood.
* Current clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances.
* Current clinically significant cardiovascular disease. Clinically significant cardiovascular disease usually includes one or more of the following: a) cardiac surgery or myocardial infarction within the last 6 months; b) unstable angina; c) coronary artery disease that required an increase in medication within the last 3 months; d) decompensated congestive heart failure; e) significant cardiac arrhythmia or conduction disturbance, particularly those resulting in a trial or ventricular fibrillation, or causing syncope, near syncope, or other alterations in mental status; f) severe mitral or aortic valvular disease; g) uncontrolled high blood pressure; h) congenital heart disease) .
* Current history of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
* Current clinically significant infectious disease, including known Acquired Immune Deficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV) infection or previous positive test for hepatitis.
* Women of childbearing potential who are not surgically sterile, not refraining from sexual activity, or not using reliable methods of contraception. Women of childbearing potential must not be pregnant (negative serum beta-hCG [human chorionic gonadotropin] at the time of screening and negative urine beta-hCG on the day of imaging) or lactating at screening. Women must avoid becoming pregnant, and must agree to refrain from sexual activity or to use reliable contraceptive methods for 30 days prior to and 30 days after administration of radiopharmaceutical imaging agents in this study. In order to participate in this study, sexually active females must be either: two or more years post-menopausal or surgically sterilized, or must be using an acceptable form of contraception (oral contraceptives for at least three months or an IUD (intrauterine device) for at least two months prior to the start of the screening visit, or various barrier methods, e.g., diaphragm or combination condom and spermicide).
* Subjects who, in the opinion of the research team, are otherwise unsuitable for a study of this type.
* Subjects who have a history of relevant severe drug allergy or hypersensitivity.
* Subjects who have received an investigational medication within the last 30 days. Additionally, the time between the last dose of the previous experimental medication and enrollment (completion of screening assessments) must be at least equal to 5 times the terminal half-life of the previous experimental medication.
* Subjects who have ever participated in an experimental study with an amyloid targeting therapy (e.g., immunotherapy, secretase inhibitor) may not be enrolled unless it can be demonstrated that the subject received only placebo in the course of the trial.
* Current clinically significant medical comorbidities, as indicated by history, physical exam, or laboratory evaluations, that might pose a potential safety risk, interfere with the absorption or metabolism of the study medication, or limit interpretation of the trial results. These include but are not limited to clinically significant hepatic, renal, pulmonary, metabolic or endocrine disease, and cancer.
* Subjects who have received a radiopharmaceutical for imaging or therapy within the past 7 days prior to the imaging session for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Florbetapir PET - change between timeframes | Year 1, Year 2-3
  The researchers will use multi-modal partial least squares (MMPLS) to integrate the volumetric MRI, tau PET, FDG PET and florbetapir PET data and investigate the potential for increased sensitivity to examine the longitudinal changes related to both brain structure and fibrillar amyloid depositions. The MMPLS based subject scores, which is free from multiple comparisons, will be the primary measure integrating information from imaging modalities. The combined primary measures will be used each to compute the number of DS or DS/AD patients in the treatment and in the placebo arms needed for a 60 month clinical trial with 80% power, two-tailed p=0.05 and assumed treatment effects of 25%. These estimated samples are indicative of each biomarker for their sensitivity.
tau PET - change between timeframes | Year 1, Year 2-3
  The researchers will use multi-modal partial least squares (MMPLS) to integrate the volumetric MRI, tau PET, FDG PET and florbetapir PET data and investigate the potential for increased sensitivity to examine the longitudinal changes related to both brain structure and fibrillar amyloid depositions. The MMPLS based subject scores, which is free from multiple comparisons, will be the primary measure integrating information from imaging modalities. The combined primary measures will be used each to compute the number of DS or DS/AD patients in the treatment and in the placebo arms needed for a 60 month clinical trial with 80% power, two-tailed p=0.05 and assumed treatment effects of 25%. These estimated samples are indicative of each biomarker for their sensitivity.
FDG PET - change between timeframes | Year 1, Year 2-3
  The researchers will use multi-modal partial least squares (MMPLS) to integrate the volumetric MRI, tau PET, FDG PET and florbetapir PET data and investigate the potential for increased sensitivity to examine the longitudinal changes related to both brain structure and fibrillar amyloid depositions. The MMPLS based subject scores, which is free from multiple comparisons, will be the primary measure integrating information from imaging modalities. The combined primary measures will be used each to compute the number of DS or DS/AD patients in the treatment and in the placebo arms needed for a 60 month clinical trial with 80% power, two-tailed p=0.05 and assumed treatment effects of 25%. These estimated samples are indicative of each biomarker for their sensitivity.
MRI - change between timeframes | Year 1, Year 2-3
  The researchers will use multi-modal partial least squares (MMPLS) to integrate the volumetric MRI, tau PET, FDG PET and florbetapir PET data and investigate the potential for increased sensitivity to examine the longitudinal changes related to both brain structure and fibrillar amyloid depositions. The MMPLS based subject scores, which is free from multiple comparisons, will be the primary measure integrating information from imaging modalities. The combined primary measures will be used each to compute the number of DS or DS/AD patients in the treatment and in the placebo arms needed for a 60 month clinical trial with 80% power, two-tailed p=0.05 and assumed treatment effects of 25%. These estimated samples are indicative of each biomarker for their sensitivity.

SECONDARY OUTCOMES:
dried blood spot collection (DBSC) analysis - change between timeframes | Year 1, Year 2-3
  (a) Detect and track RNA biomarkers longitudinally from a single dried blood spot (DBS) using next generation RNA sequencing (RNA-Seq) in prospectively assessed DS, DS/AD and NC, (b) Study and identify biomarkers with the greatest rate of change in DS patients who are at differential risk levels for the development of AD dementia, and (c) Correlate the RNA biomarkers with imaging (FDG-PET, FBP (Florbetapir F18)-PET, MRI, tau PET) that are concurrently being gathered in the proposed study populations.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan N Sabbagh, MD, Principal Investigator — Barrow Neurological Institute
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No